CLINICAL TRIAL: NCT01975168
Title: The Effect Evaluation of Laser Acupuncture in Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Cheng-Che Lin, Doctor of Chinese Medicine Department, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: KMUH-LAAC-OB-001
Record Dates: First submitted 2013-10-23; First posted 2013-11-04 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Obesity
Keywords: laser acupuncture; obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): arrange laser acupuncture intervention for 12 weeks, then cross over to sham laser acupuncture intervention for 12 weeks
  Interventions: Device: Handylaser Trion laser acupuncture
- Group 2 (Sham Comparator): arrange sham laser acupuncture for 12 weeks, then cross over to laser acupuncture for 12 weeks
  Interventions: Device: Handylaser Trion laser acupuncture

INTERVENTIONS:
Device: Handylaser Trion laser acupuncture — intervention interval is 3 times per week for 12 weeks
  Other Names: Handylaser Trion

SUMMARY:
A randomized double-blind placebo-controlled crossover trial is conducted. 200 subjects aged above 20 years with body mass index (BMI) more than 25 kg/m2 are randomly divided into 2 groups (Group 1 and Group 2). Group 1 receives laser acupuncture therapy first while Group 2 receives sham laser acupuncture therapy first. After 12 weeks of treatment and 14 days of washout, Group 1 switch to sham laser acupuncture therapy while Group 2 switch to laser acupuncture for 12 weeks. The subjects are treated with a gallium aluminum arsenide Handylaser Trion, which is used to apply at each of the acupuncture points for 10 seconds every time, 3 times per week. The measurements of outcomes are performed in the beginning, weekly during treatment, and monthly after treatment for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index over 25 kg/m2 or Waist girth over 80cm in female, waist girth over 90cm in male

Exclusion Criteria:

* Pathmakers user
* Epilepsy history
* Pregnancy
* Immuno-inhibiting agents user
* Malignancy
* Skin contacted disease
* Weight controlled agents user during trial period
* Eating disorder

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
body composition | 12 weeks
  body weight

SECONDARY OUTCOMES:
body mass index | 12 weeks

OTHER OUTCOMES:
waist circumference | 12 weeks
hip circumference | 12 weeks
body fat | 12 weeks
blood pressure | 12 weeks
heart rate | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Che Lin, MD, Study Chair — Doctor of Chinese Medicine Department, Kaohsiung Medical University Hospital; Hung-Yi Chuang, ScD, MD, Study Director — Department of Public Health, College of Health Sciences, Kaohsiung Medical University; Chen-Cheng Yang, MD, Principal Investigator — Family Medicine Department, Kaohsiung Medical University Hospital and Kaohsiung Municipal Ta-Tung Hospital
Locations (1):
- Chinese Medicine Department Clinic, Kaohsiung Medical University, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Wozniak P, Stachowiak G, Pieta-Dolinska A, Oszukowski P. Laser acupuncture and low-calorie diet during visceral obesity therapy after menopause. Acta Obstet Gynecol Scand. 2003 Jan;82(1):69-73. doi: 10.1034/j.1600-0412.2003.820113.x. PMID 12580844